CLINICAL TRIAL: NCT05004753
Title: A Prospective, Randomized, Multi-center, Open Label, Interventional Study to Evaluate the Safety and Efficacy of Artemisinin 500 mg Capsule in Treatment of Adult Subjects With COVID-19
Brief Title: A Study to Evaluate the Safety and Efficacy of Artemisinin- a Herbal Supplement on COVID-19 Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Collaborators: Windlas Biotech Private Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTI/WBPL/P4/2020/01
Record Dates: First submitted 2021-07-26; First posted 2021-08-13 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — artemisinin; Dexamethasone

STUDY DESIGN:
Intervention Model Description: 2 to 1 ratio
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artemisinin 500mg (Experimental): The dose regimen will be in cycles. In a cycle a subject will receive Artemisinin 500 mg capsule once daily plus SOC on Day 1 to Day 5 followed by 5 days off (no dosing of Artemisinin) or SOC alone. A subject can have a total of consecutive 3 cycles maximum. Here SOC is Standard of Care as per CLINICAL MANAGEMENT PROTOCOL: COVID-19, Government of India Ministry of Health and Family Welfare Directorate General of Health Services (EMR Division)
  Interventions: Dietary Supplement: Artemisinin
- Standard of Care (Active Comparator): Standard of Care as per CLINICAL MANAGEMENT PROTOCOL: COVID-19, Government of India Ministry of Health and Family Welfare Directorate General of Health Services (EMR Division) Mild Patients: HYDROXYCHLOROQUINE Moderate Patients: Dexamethasone - OD for 05
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Dietary Supplement: Artemisinin — a herbal supplement
  Arms: Artemisinin 500mg
Drug: Dexamethasone — corticosteroids
  Arms: Standard of Care

SUMMARY:
This will be an open label, prospective, multi-center, comparative, interventional study to evaluate safety and efficacy of Artemisinin 500 mg in subjects with mild to moderate COVID-19. Initially subjects having mild to moderate COVID-19 will be screened as per predefined eligibility criteria for the study. Eligible 120 subjects will be enrolled to receive treatment with Artemisinin and SOC (Standard of Care as per CLINICAL MANAGEMENT PROTOCOL: COVID-19, Government of India Ministry of Health and Family Welfare Directorate General of Health Services (EMR Division)) or SOC. Subjects will be randomized in 2:1 ratio. Group 1 will have 80 subjects and Group 2 will have 40 subjects.

DETAILED DESCRIPTION:
The study will involve screening (Day 1), treatment period of up to maximum 28 days till end of study. The investigator shall make every effort to follow the schedule of study assessments and procedures. A window period of 1 day will be allowed for assessments post randomization. Screening Upon obtaining the written informed consent the subjects will be screened to confirm the eligibility for participating in this study. If RT PCR result is available for the subject then screening and baseline (randomization) activity will be on the same day. As per the Investigator discretion, the subjects meeting the criteria will be hospitalized for the first cycle of treatment Treatment period Subjects will receive investigational product and SOC after randomization as per protocol. Subject's compliance with the study treatment regimen of Artemisinin one (1) capsule a day for five (5) days, will be assessed during treatment period. Subjects receiving at least one dose of study treatment will be included in the safety analysis. Efficacy analysis will be conducted in completers (subjects who have completed at least 5 consecutive days of dosing in either arm) The first cycle of the study drug treatment will be given in the hospital, for which the subjects have to be hospitalized till Day 5, unless prolongation of hospital stay is necessary as per the investigator. On day 14, telephonic follow up is done for subjects discharged after Day 5. For Day 28 visit all subjects will visit the hospital to complete the End of Study activities.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of ≥18 to 60 years of age both inclusive
2. Subjects willing to give informed consent and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
3. Confirmed case of COVID-19 infection by RT-PCR and mild and moderate (without oxygen therapy or assisted ventilation) cases of COVID-19. Scores of 2-4 on the WHO Clinical Progression Scale
4. Time interval between symptoms onset and randomization of no more than 7 days
5. One or more of the following symptoms:

   Fever Cough Sore throat Headache Nasal congestion Malaise Diarrhea Loss of smell Loss of taste
6. Male and female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

Exclusion Criteria:

1. Subjects with history of severe infections (pneumonia, septicemia, etc.), severe cardiac or pulmonary diseases, or received immunosuppressive therapy or other investigational drugs within the previous 30 days of screening
2. Known or suspected hypersensitivity to Artemisinin
3. Women of child bearing potential who are currently pregnant, lactating or who are not willing to use contraception during the entire duration of the study
4. Men who are unwilling to use contraception while receiving investigational product
5. Subjects with history of severe disease other than COVID-19 which is expected to prevent compliance with the present protocol
6. Subjects with history of severe renal and hepatic impairment. (creatine ≥2 mg/dl; liver enzymes and bilirubin 2.5 times ULN; alkaline phosphatase 1.5 times ULN)
7. Recent treatment with Artemisinin or Artemisinin based antimalarials in the past 7 days
8. Known history of failure to control systemic fungal, bacterial or viral infection
9. Patients with the history of following co-morbidities: diabetes, hypertension with or without cardiac symptoms, morbid obesity with diabetes and/or hypertension or any other metabolic syndrome
10. Subjects with known human immunodeficiency virus (HIV) or hepatitis B or C classes of active viral infection
11. Have a history of neurological or psychiatric disorders, including epilepsy or dementia
12. Subjects for whom ventilator support is required at screening
13. Patients not willing to stay in hospital for 5 days of isolation following diagnosis of Covid-19
14. Subjects not willing to give their informed consent to participate in the clinical trial
15. According to the investigator judgment there are concomitant diseases with a serious safety hazard or affect the subject
16. Using other experimental drugs or participating in other clinical trials in the prior one month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Safety Assessments | 28 days
  * Incidence of adverse events during the study.
  * Incidence of serious adverse events during the study.

SECONDARY OUTCOMES:
Efficacy Assessments | 28 days
  * Improvement rate in severity of COVID-19 per 8-point WHO COVID-19 Clinical Improvement Ordinal Scale.
  * Improvement rate in severity of COVID-19 per the Duration of Symptoms.
  Clinical improvement is defined as
  • A rate decrease to categories 1, 2, 3, or 4.

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Kumar, Study Chair — Windlas Biotech Private Limited
Locations (3):
- India (3):
  - Government Medical College & Government General Hospital, Srikakulam, Srikakulam, Andhra Pradesh
  - Rajarshi Chhatrapati Shahu Maharaj Government Medical college and Chhatrapati Pramila Raje Hospital, Kolhāpur, Maharashtra
  - Seven Star Hospital, Nagpur, Maharashtra

REFERENCES:
- [Result] Trieu V, Saund S, Rahate PV, Barge VB, Nalk KS, Windlass H, Uckun FM. Targeting TGF-beta pathway with COVID-19 Drug Candidate ARTIVeda/PulmoHeal Accelerates Recovery from Mild-Moderate COVID-19. Clinical Investigation (2021) 11(1), 10-18